CLINICAL TRIAL: NCT04241250
Title: Transspinal Versus Epidural Stimulation for Exoskeletal Assisted Walking After Spinal Cord Injury
Brief Title: Neuromodulation Techniques After SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B3456-P
Record Dates: First submitted 2020-01-10; First posted 2020-01-27 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Spinal Cord Injury
Keywords: Robotic Exoskeleton; Epidural Stimulation; Transspinal stimulation; Spinal cord injury; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Exoskeletal assisted walking and spinal cord epidural stimulation (EAW+SCES) Exoskeletal assisted walking and Transspinal stimulation (EAW+TS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- EAW+SCES (Experimental): Three months of exoskeleton training followed by 6 months of epidural stimulation.
  Interventions: Device: EAW+SCES (exoskelton and spinal cord epidural stimulation)
- EAW+TS (Experimental): Three months of exoskeleton training followed by 6 months of transspinal stimulation.
  Interventions: Device: EAW+TS (exoskelton and transspinal stimulation)

INTERVENTIONS:
Device: EAW+SCES (exoskelton and spinal cord epidural stimulation) — Three months of exoskeleton training followed by 6 months of epidural stimulation.
  Arms: EAW+SCES
Device: EAW+TS (exoskelton and transspinal stimulation) — Three months of exoskeleton training followed by 6 months of transspinal stimulation.
  Arms: EAW+TS

SUMMARY:
Spinal cord injury (SCI) leads to several health-related consequences often linked to reduced levels of physical activity. Direct stimulation of the spinal cord, either through implanted devices or surface stimulation, has been combined with intense physical therapy assisted treadmill walking to facilitate independent standing and stepping. These current methods require 3-4 highly skilled therapists and may not be feasible in all rehabilitation settings, especially when considering the growing number of SCI patients each year. Therefore, the use of robotic exoskeleton suits combined with direct stimulation of the spinal cord (requiring 1-2 therapists) may offer an alternative rehabilitation approach to overcome their limited abilities to stand and walk. Such improvements may also help to reverse or eliminate other health-related consequences associated with SCI. The pilot work will provide the preliminary evidence required to design future clinical trials for Veterans and civilians with SCI to restore overground mobility.

DETAILED DESCRIPTION:
Restoring locomotion following spinal cord injury (SCI) has been the focus of years of research aimed at ameliorating several of health-related comorbidities. Spinal cord epidural stimulation (SCES) exhibits the rehabilitation potential of restoring locomotion in individuals with SCI when combined with intensive locomotion training. Despite this potential, such protocols are likely impractical when applied across large clinical SCI populations due to high monetary costs. Similar to SCES, transspinal stimulation (TS) has also exhibited neuromodulatory benefits by externally stimulating lumbro-sacral neural circuity to generate step-like activities in persons with complete SCI; however, these techniques also require intense gait training. Recently robotic exoskeletons have been used as a promising tool to circumvent limitations associated with labor-intensive locomotor training, and have been safely used as an effective approach in improving levels of physical activity in persons with complete SCI.

Recent work has demonstrated the benefits of combining EAW and neuromodulatory techniques. Following 12-weeks of EAW+SCES training, improvements in locomotion led researchers to decrease the amount of EAW swing assistance to 35% in a person with a C7 complete SCI. This was accompanied by 573 unassisted steps, which represents 50% of the total number of steps taken during that session. Electromyographic (EMG) activity also increased during both stance and swing phases, reflecting the individual's ability to rhythmically fire paralyzed muscles during EAW+SCES. Additionally, cardio-metabolic loads were increased during exoskeletal stepping when combined with SCES as compared to stepping without SCES. The participant also showed a modest decrease in his total and regional absolute fat mass. These preliminary findings suggest that neuromodulation using SCES with exoskeletal ambulation may provide a feasible rehabilitation approach for persons with SCI. The goal of the current study is to examine and compare the effects of EAW combined with SCES or TS in persons with motor complete SCI. The data generated from this application will also enable larger clinal trials to explore ways to optimize exoskeletal assisted gait training through the use of different neuromodulation modalities with SCI.

Following a repeated-measure design, 10 participants with chronic, motor complete (AIS A and B) SCI (age:18-60 years) will be randomly assigned to participate in either 6-months of EAW+SCES (n=5) or EAW+TS (n=5) training. The entire duration of the trial will be approximately 1 year for each participant. Initially, participants will undergo 3-months of EAW training (3 sessions/week), which will be followed by randomization into either a EAW+SCES group or EAW+TS group for an additional 6-months of training (both groups: 3 sessions/week) and a 3-month follow-up period for both groups. Measurements at baseline (BL: prior to EAW) and 4 post-intervention timepoints will occur every 3-months (P1: following 3-months of EAW; P2: following 3-months of EAW+TS or EAW+SCES; P3: after completing 6-months of EAW+TS or EAW+SCES; P4: 3-months after termination of EAW+TS or EAW+SCES).

This pilot work will have 3 specific aims: Aim 1. The investigators will determine and compare improvements to locomotor control following 6 months of EAW+TS and EAW+SCES as measured by 10-meter walking speed, the number of unassisted EAW steps, and EMG activity.

Aim 2. The investigators will determine and compare improvements to cardio-metabolic risk factors following 6 months of EAW+TS and EAW+SCES as measured by total and regional body composition, oxygen uptake, and fasting lipid profile.

Aim 3. The investigators will determine and compare improvements in bladder health following 6 months of EAW+TS and EAW+SCES as measured by bladder filling and emptying

ELIGIBILITY:
Inclusion Criteria:

* All participants will be between 18-70 years old, male, with traumatic motor complete SCI and level of injury of T10 and above, as determined by EMG testing and International Standards for Neurological Classification of SCI (ISNCSCI) exam
* All participants will undergo ISNCSCI examination for neurological level and function and only those with American Spinal Injury Classification (AIS A and B; i.e. motor deficit below the level of injury) will be included

Exclusion Criteria:

Participants with any of the following pre-existing medical conditions will be excluded from the current trial:

* Diagnosis of neurological injury other than SCI, including cauda equina or distal conus injuries resulting in limb or sacral areflexia
* Unhealed fracture in either lower or upper extremities
* Severe scoliosis, hip knee range of motion (ROM) or flexion knee contractures preventing positioning in an exoskeleton or plantarflexion contracture greater than 20 degrees
* Untreated or uncontrolled hypertension defined as high resting blood pressure greater than 140/90 mmHg and severe orthostatic hypotension (drop greater than 20 mmHg compared to resting supine blood pressure) or incapable to maintain a sitting or EAW standing posture
* Other medical conditions including cardiovascular disease, uncontrolled type II DM, uncontrolled hypertension, and those on insulin, pressures sores stage 3 or greater, or symptomatic urinary tract infection
* Unable to fit in the device for any reason
* Taking anti-coagulants or anti-platelet agents, including aspirin if unable to be off this medication for medical reasons
* Implanted pacemakers and/or implanted defibrillator devices
* DXA T-Score less than -2.5. Scans done will include total body, dual hips and knees. Total hip BMD T-scores < -3.5 and knee BMD scores of less than 0.6 g/cm2
* Functional upper and lower extremity ROM, strength, spasticity and skin integrity will also have assessed prior to enrollment in the program.

  * The Modified Ashworth Scale will be used to ensure safety of the participants prior to engagement in the rehabilitation program

    * Participants with severe spasticity or limited ROM will be excluded from the trial
    * This is based on the Ekso manufacturer's recommendations
* Untreatable severe spasticity judged to be contraindicated by the site Physician
* Pressure ulcer of the trunk, pelvic area, or lower extremities of grade 3 or more
* Psychopathology documentation in the medical record or history that may conflict with study objectives
* Any condition that, in the judgment of the principal investigator or medical provider, precludes safe participation in the study and/or increases the risk of infection

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
10-meter walking speed (m/sec) | 9 months
  After fitted in the robotic exoskeleton, the participant will be asked to walk for 10-meter distance and the time and speed will be determined.
Muscles electromyography (EMG) activity (micro-volts) | 9 months
  EMG activity will measure electrical activity from 12 leg muscles of hip, knee, and ankle joints during locomotion

SECONDARY OUTCOMES:
Fat mass and fat-free mass (kg) | 9 months
  Body composition will be captured using dual energy x-ray absorptiometry (DXA) to measure fat mass (kg) and fat-free mass (kg) every 3 months during the course of the trial.
Oxygen Uptake (ml/min) | 9 months
  Oxygen uptake during resting, standing and walking will be measured during 6 minutes walking test every 3 months during the course of the trial.
Fasting lipid profile (mg/dl) | 9 months
  After overnight fast, blood will be drawn to measure your circulating triglycerides, low and high density lipoproteins and cholesterol.

OTHER OUTCOMES:
Volume of bladder Capacity during filling and voiding (ml) | 9 months
  A multichannel urodynamics system (Laborie) will be used to perform urodynamic studies . A urethral catheter will be placed, and saline is infused into the bladder. A pressure transducer is also inserted into the bladder and records pressure during filling. We will then measure the volume of the bladder during filling and during emptying.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Gorgey, PhD PT, Principal Investigator — Hunter Holmes McGuire VA Medical Center, Richmond, VA
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hachmann JT, Yousak A, Wallner JJ, Gad PN, Edgerton VR, Gorgey AS. Epidural spinal cord stimulation as an intervention for motor recovery after motor complete spinal cord injury. J Neurophysiol. 2021 Dec 1;126(6):1843-1859. doi: 10.1152/jn.00020.2021. Epub 2021 Oct 20. PMID 34669485
- [Result] Gorgey AS, Trainer R, Sutor TW, Goldsmith JA, Alazzam A, Goetz LL, Lester D, Lavis TD. A case study of percutaneous epidural stimulation to enable motor control in two men after spinal cord injury. Nat Commun. 2023 Apr 12;14(1):2064. doi: 10.1038/s41467-023-37845-7. PMID 37045845
- [Result] Alazzam AM, Ballance WB, Smith AC, Rejc E, Weber KA 2nd, Trainer R, Gorgey AS. Peak Slope Ratio of the Recruitment Curves Compared to Muscle Evoked Potentials to Optimize Standing Configurations with Percutaneous Epidural Stimulation after Spinal Cord Injury. J Clin Med. 2024 Feb 27;13(5):1344. doi: 10.3390/jcm13051344. PMID 38592158
- [Result] Gorgey AS, Goldsmith J, Alazzam A, Trainer R. Effects of percutaneously-implanted epidural stimulation on cardiovascular autonomic function and spasticity after complete spinal cord injury: A case report. Front Neurosci. 2023 Feb 16;17:1112853. doi: 10.3389/fnins.2023.1112853. eCollection 2023. PMID 36875669

DOCUMENTS (1):
  • Informed Consent Form (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT04241250/ICF_000.pdf